CLINICAL TRIAL: NCT06231316
Title: Preventing Spinal Hypotension During Cesarean Birth With Two Initial Boluses of Norepinephrine
Brief Title: Preventing Hypotension in the Spine During Cesarean Delivery.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Mousa Abd Elsadek Ahmed, Doctor, Assiut University
Other Study IDs: PSHDCB
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Norepinephrine Injection — Norepinephrine is both a neurotransmitter and a hormone. It is essential vasopressor for rapid blood pressure support, crucial in maintaining hemodynamic stability

SUMMARY:
Examining the advantages associated with the utilization of noradrenaline in preventing spinal hypotension during cesarean births. This involves assessing the positive outcomes and potential benefits derived from incorporating noradrenaline into the medical approach.

DETAILED DESCRIPTION:
Spinal anesthesia is used during cesarean section to provide rapid onset and dense block of motor and sensory nerves, intraoperative analgesia, and help patients remain conscious (1,2).Hypotension is common during induction of spinal anesthesia for cesarean delivery (CD) (3).If not promptly treated, a decrease in blood pressure (BP) can have deleterious effects, which include maternal nausea, vomiting, dizziness, and cardiovascular instability as well as decreased uteroplacental blood flow with resultant fetal acidosis, hypoxia, and bradycardia.In the last decade, the α-agonist phenylephrine (PE) has been the vasopressor of choice for the prevention and treatment of spinal induced hypotension (4).To prevent and treat postspinal anesthesia hypotension during cesarean section, vasopressors are recommended. Vasopressors (especially potent α-adrenergic receptor agonists) help offset the decrease in arteriolar dilation and peripheral vascular resistance caused by sympathetic nerve blockade after spinal anesthesia and may be associated with decreased incidence of neonatal acidosis.(5,6). Norepinephrine is another vasopressor that was recently introduced in obstetric anesthesia (7). Norepinephrine is characterized by α-adrenergic agonistic activity in addition to a weak β-adrenergic agonistic activity; thus, norepinephrine is considered a vasopressor with minimal cardiac depressant effect(7).; these pharmacologic properties would make norepinephrine an attractive alternative to phenylephrine and ephedrine in obstetric anesthesia. Although the use of norepinephrine for prophylaxis against postspinal hypotension has shown promising results,(7,8) evidence is lacking on the optimum dose for norepinephrine infusion during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* The subject is scheduled for elective cesarean section .
* No obvious abnormalities in preoperative ECG, blood routine, electrolytes, and other tests.
* ASA class 1-3.

Exclusion Criteria:

* Patients have body mass index (BMI) >35 kg/m2. -Patients are known hypersensitivity to any of the drugs that would be used in the study. -
* Severe cardiac, renal, lung, or liver diseases.
* Eclampsia or preexisting hypertension (baseline systolic blood pressure ≥160 mmHg)
* hemoglobin <7 g/dL, or fetal distress.
* Patients that are immunologically compromised.
* Sleep apnea syndrome or difficult airway. 8.preexisting hypoxemia (Spo2< 90 %).
* Patient refusal.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Sample size was calculated using Epi- Info7. Based on Frequency of spinal hypotension decrease to 20% in patients received0.5_.10mg epinephrine ( put ref . ). With a confidence limits 5% and a confidence level of 90% the minimum patients required for this study is 173cases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of postspinal hypotension | baseline
  Assessment of how often blood pressure decreases following spinal anesthesia, crucial for proactive management in medical procedures.

SECONDARY OUTCOMES:
Hemodynamic data | baseline
  the frequency of severe postspinal hypotension, frequency of postdelivery hypotension (defined as decreased SBP less than 80% of the baseline reading after delivery of the fetus and starting oxytocin infusion), frequency of intraoperative nausea and vomiting, frequency of intraoperative hypertension.

REFERENCES:
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] Sakata K, Yoshimura N, Tanabe K, Kito K, Nagase K, Iida H. Prediction of hypotension during spinal anesthesia for elective cesarean section by altered heart rate variability induced by postural change. Int J Obstet Anesth. 2017 Feb;29:34-38. doi: 10.1016/j.ijoa.2016.09.004. Epub 2016 Sep 22. PMID 27789074
- [Background] Kuhn JC, Hauge TH, Rosseland LA, Dahl V, Langesaeter E. Hemodynamics of Phenylephrine Infusion Versus Lower Extremity Compression During Spinal Anesthesia for Cesarean Delivery: A Randomized, Double-Blind, Placebo-Controlled Study. Anesth Analg. 2016 Apr;122(4):1120-9. doi: 10.1213/ANE.0000000000001174. PMID 26991619
- [Background] Macarthur A, Riley ET. Obstetric anesthesia controversies: vasopressor choice for postspinal hypotension during cesarean delivery. Int Anesthesiol Clin. 2007 Winter;45(1):115-32. doi: 10.1097/AIA.0b013e31802b8d53. No abstract available. PMID 17215703
- [Background] Lee JE, George RB, Habib AS. Spinal-induced hypotension: Incidence, mechanisms, prophylaxis, and management: Summarizing 20 years of research. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):57-68. doi: 10.1016/j.bpa.2017.01.001. Epub 2017 Jan 8. PMID 28625306
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852